CLINICAL TRIAL: NCT03479008
Title: Testing of a New Therapeutic Vibration Device to Reduce Neuromuscular Weakness in Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Benjamin Bassin, Professor in the Department of Emergency Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00129402
Record Dates: First submitted 2018-02-28; First posted 2018-03-27 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Critically Ill; Post Intensive Care Syndrome
MeSH Terms: conditions — Critical Illness; postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Healthy volunteers (iterative device development) (Other): This phase will recruit healthy volunteers who will be vibrated with the prototype device using various vibration frequencies to determine which frequency produces the optimal physiologic response. Physiologic responses will be determined with a number of devices capable of measuring such things as tissue oxygenation, oxygen consumption, and muscle activity. Volunteers will be randomized to receive alternating 5 minute episodes of various vibration frequencies.
  Interventions: Diagnostic Test: Therapeutic Vibration Device

INTERVENTIONS:
Diagnostic Test: Therapeutic Vibration Device — The Therapeutic Vibration Device is capable of applying force through the axial skeletal spine, through bidirectional compression loading (or prestressing) between the shoulder and the plantar surfaces of the feet. It is placed around the body like a mobile frame so that the applied vibration can affect the whole body. The vibration actuators (drivers) are mobile and can vary in size, frequency response, and force. The design minimizes the possibility of mechanical interference for ventilated/intubated patients.

SUMMARY:
Objective: Test the ability of vibration to produce physiologic, biochemical, and anatomic changes consistent with exercise that would help prevent the development of muscle weakness that occurs when patients are immobile for long periods of time.

DETAILED DESCRIPTION:
During critical illness, patients who are immobilized for more than a few days develop severe muscle and nerve weakness despite receiving full supportive care, which may include physical therapy. In patients requiring mechanical ventilation (a device that breaths for them) for longer than 7 days, the incidence of ICU-acquired weakness is reported to be between 25% and 60%. Such weakness may contribute to increased duration of mechanical ventilation, increased length of stay in the ICU and hospital, and poor quality of life among survivors. This is part of the newly recognized Post Intensive Care Syndrome (PICS). Moreover, patients who are transferred from the ICU to a high-dependency unit (HDU), intensive therapy unit (ITU), post-operative therapy or outpatient ambulatory care need to be mobile as well as awake for any physical therapy. Patients affected by sepsis (severe blood stream infections), osteoarthritis, spinal cord injury, stroke, multiple sclerosis, cerebral palsy, cancer, and other illnesses suffer muscle loss and weakness. Early mobilization (EM) has demonstrated the ability to significantly reduce the detrimental effects of prolonged immobilization such as polyneuropathy and myopathy (nerve damage and muscle weakness), which in turn reduces the time patients spend on mechanical ventilation and the overall length of hospital stay. EM treatments include intense physical therapy, cycle ergometry, transcutaneous electrical muscle stimulation (TEMS) and continuous lateral rotational therapy (CLRT). However, carrying out intense physical therapy using therapists is impractical (especially at smaller hospitals) and cannot be implemented in heavily sedated patients (patients who cannot cooperate). Evidence suggests that vibration may be capable of producing adequate muscle contraction via muscle-spinal loops that may be sufficient to reduce or prevent nerve damage and muscle weakness caused by prolonged immobilization thus serving as an effective treatment making patients stronger when they leave the ICU.

The purpose of this study is to test a prototype vibration device and strategy on its ability to exercise large muscle groups, increase muscle blood flow, and increase circulating levels of blood chemicals associated with exercise/activity. The study will be used to find optimal vibration frequencies that provide maximal evidence of associated muscle activity. Eventually the investigators hope to see a vibration device capable of delivering a more effective therapy compared to the smaller gains derived from traditional measures of physical therapy in critically ill patients such as TEMS, CLRT and cycle ergometry to patients. The vibration device may directly benefit the patient in terms of health, length of stay and reduced re-admission, hospital staff in terms of productivity (i.e., through reduction in nursing effort) and the hospital in terms of reduced cost and return on investment. Its value is also envisioned in many other populations of immobilized acutely ill and injured patients as well as those with chronic conditions.

Originally registered as a single record, this registration has been simplified to clarify the outcomes measured from the work with healthy volunteers. A new registration which will include the relevant outcomes for the trial part that will enroll hospitalized participants will be registered prior to their enrollment. The current registration will remain open until it is certain that no additional modifications of the device are required to go through a new round of iterative testing with healthy volunteers. While the total number of participants to be enrolled is larger than some early feasibility trials, the testing is done in small iterative batches to determine whether additional design changes are required. Each of these is generally less than 10 individuals.

ELIGIBILITY:
Exclusion Criteria:

1. Known pregnancy
2. Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Bassin, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saxena H, Ward KR, Krishnan C, Epureanu BI. Effect of Multi-Frequency Whole-Body Vibration on Muscle Activation, Metabolic Cost and Regional Tissue Oxygenation. IEEE Access. 2020;8:140445-140455. doi: 10.1109/access.2020.3011691. Epub 2020 Jul 24. PMID 34036017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to actual testing for the outcomes listed in this registration, 8 participants were recruited and consented for tuning and characterizing the device prior to structured testing.
Pre-assignment Details: 6 participants consented for testing the device did not come in for their first appointment.
Groups:
- Healthy Volunteers (Iterative Device Development): This phase recruited healthy volunteers who were be vibrated with the prototype device using various vibration frequencies to determine which frequency produces the optimal physiologic response. Physiologic responses were determined with a number of devices capable of measuring such things as tissue oxygenation, oxygen consumption, and muscle activity. Volunteers were randomized to receive alternating 5 minute episodes of various vibration frequencies.
  Therapeutic Vibration Device: The Therapeutic Vibration Device is capable of applying force through the axial skeletal spine, through bidirectional compression loading (or prestressing) between the shoulder and the plantar surfaces of the feet. It is placed around the body like a mobile frame so that the applied vibration can affect the whole body. The vibration actuators (drivers) are mobile and can vary in size, frequency response, and force. The design minimizes the possibility of mechanical interference for ventilated/intubated patients.
Period: Overall Study
Arm/Group | Healthy Volunteers (Iterative Device Development)
Started | 22
Completed | 19
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers (Iterative Device Development)
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Regional Hemoglobin Oxygen Saturation
Description: Change in tissue regional hemoglobin oxygen saturation (rSO2) using near infrared spectroscopy of the thighs,calf, and biceps Baseline measurements were taken for 1 minute and vibration period was for 10 minutes.
  The mean value of rSO2 for 1 minute preceding vibration was computed as the baseline value. For the data collected during vibration, a moving average peak analysis for every 1 minute for 10 minutes of rSO2 data was carried out. The maximum value of the moving average was selected as the mean value of vibration. The moving average peak analysis was independently conducted for all three measurements from GL, RF and BB.
Time Frame: 10 minutes
Population: One dataset was discarded due to poor data quality due to instrumentation issues encountered during testing.
Measure: Mean (Standard Error); unit: percent of oxygenation
Groups:
- Healthy Volunteers (1st Iteration of Device Development): This phase recruited healthy volunteers who were be vibrated with the prototype device using various vibration frequencies to determine which frequency produces the optimal physiologic response. Physiologic responses were determined with a number of devices capable of measuring such things as tissue oxygenation, oxygen consumption, and muscle activity. Volunteers were randomized to receive alternating 5 minute episodes of various vibration frequencies.
  Therapeutic Vibration Device: The Therapeutic Vibration Device is capable of applying force through the axial skeletal spine, through bidirectional compression loading (or prestressing) between the shoulder and the plantar surfaces of the feet. It is placed around the body like a mobile frame so that the applied vibration can affect the whole body. The vibration actuators (drivers) are mobile and can vary in size, frequency response, and force. The design minimizes the possibility of mechanical interference for ventilated/intubated patients.
Arm/Group | Healthy Volunteers (1st Iteration of Device Development)
Number analyzed (Participants) | 18
percent of oxygenation
  Thighs (baseline) | 75.65 (0.98)
  Thighs (during stimulation | 77.01 (1.09)
  Calf muscle (baseline) | 73.83 (0.93)
  Calf (during stimulation) | 77.09 (1.13)
  Biceps (baseline) | 72.23 (1.27)
  Biceps (during stimulation) | 74.15 (1.40)
Statistical Analysis 1: Comparison: Healthy Volunteers (1st Iteration of Device Development); This presents the p value for the thigh comparison baseline to during stimulation; Test type: Other; p < 0.0001, ANOVA — Statistical significance level was set at p <0.05 for all tests
Statistical Analysis 2: Comparison: Healthy Volunteers (1st Iteration of Device Development); This presents the p value for the calf comparisons between baseline and during stimulation; Test type: Superiority; p < 0.0001, ANOVA — Statistical significance level was set at p < 0.05 for all tests
Statistical Analysis 3: Comparison: Healthy Volunteers (1st Iteration of Device Development); This statistical analysis presents the data for the biceps comparisons between baseline and during stimulation; Test type: Other; p < 0.001, ANOVA — Statistical significance level was set at p < 0.05 for all tests

2. Primary Outcome: VO2 and VCO2
Description: Oxygen consumption using a VO2 monitor and mask For the baseline data, a mean of 3 minutes of the segment preceding vibration was computed. For the data collected during vibration, a moving average peak analysis for every 3 minutes for 10 minutes of VO2, VCO2 data was carried out. The maximum value of the moving average was selected as the mean value. This methodology of segment extraction precluded the possibility of picking up short transient changes in metabolic data and helped ensure selection of steady set of values of metabolic variables which estimated the true response of the participant.
Time Frame: baseline and during device use (10 minutes)
Population: Three datasets were discarded due to poor data quality due to instrumentation issues encountered during testing.
Measure: Mean (Standard Error); unit: ml/(kg*min)
Groups:
- Healthy Volunteers (1st Iteration of Device Development): This phase recruited healthy volunteers who were vibrated with the prototype device using various vibration frequencies to determine which frequency produces the optimal physiologic response. Physiologic responses were determined with a number of devices capable of measuring such things as tissue oxygenation, oxygen consumption, and muscle activity. Volunteers were randomized to receive alternating 5 minute episodes of various vibration frequencies.
  Therapeutic Vibration Device: The Therapeutic Vibration Device is capable of applying force through the axial skeletal spine, through bidirectional compression loading (or prestressing) between the shoulder and the plantar surfaces of the feet. It is placed around the body like a mobile frame so that the applied vibration can affect the whole body. The vibration actuators (drivers) are mobile and can vary in size, frequency response, and force. The design minimizes the possibility of mechanical interference for ventilated/intubated patients.
Arm/Group | Healthy Volunteers (1st Iteration of Device Development)
Number analyzed (Participants) | 16
ml/(kg*min)
  VO2 (baseline) | 3.19 (0.16)
  VO2 (during stimulation) | 3.84 (.22)
  VCO2 (baseline) | 2.54 (.14)
  VCO2 (during stimulation) | 3.07 (0.18)
Statistical Analysis 1: Comparison: Healthy Volunteers (1st Iteration of Device Development); The P value below applies to the VO2; Test type: Superiority; p < 0.0001, post-hoc analysis; with Bonferroni correction
Statistical Analysis 2: Comparison: Healthy Volunteers (1st Iteration of Device Development); This p value applies to the VCO2; Test type: Superiority; p < 0.001, post-hoc analysis; with Bonferroni correction

3. Primary Outcome: Energy Expenditure
Description: For the baseline data, a mean of 3 minutes of the segment preceding vibration was computed. For the data collected during vibration, a moving average peak analysis for every 3 minutes for 10 minutes of EE data was carried out. The maximum value of the moving average was selected as the mean value. This methodology of segment extraction precluded the possibility of picking up short transient changes in metabolic data and helped ensure selection of steady set of values of metabolic variables which estimated the true response of the participant.
Time Frame: 10 minutes
Population: Three datasets were discarded due to poor data quality due to instrumentation issues encountered during testing.
Measure: Mean (Standard Error); unit: kcal/minute
Arm/Group | Healthy Volunteers (1st Iteration of Device Development)
Number analyzed (Participants) | 16
kcal/minute
  Baseline | 1.12 (0.07)
  Vibration | 1.35 (0.09)
Statistical Analysis 1: Comparison: Healthy Volunteers (1st Iteration of Device Development); Test type: Superiority; p < 0.0001, post-hoc analysis; with Bonferroni correction

4. Primary Outcome: Minute Variation
Description: For the baseline data, a mean of 3 minutes of the segment preceding vibration was computed. For the data collected during vibration, a moving average peak analysis for every 3 minutes for 10 minutes of data was carried out. The maximum value of the moving average was selected as the mean value. This methodology of segment extraction precluded the possibility of picking up short transient changes in metabolic data and helped ensure selection of steady set of values of metabolic variables which estimated the true response of the participant.
Time Frame: 10 minutes
Population: Three datasets were discarded due to poor data quality due to instrumentation issues encountered during testing.
Measure: Mean (Standard Error); unit: liters/minute
Arm/Group | Healthy Volunteers (1st Iteration of Device Development)
Number analyzed (Participants) | 16
liters/minute
  Baseline | 7.09 (0.40)
  Vibration | 8.50 (0.55)
Statistical Analysis 1: Comparison: Healthy Volunteers (1st Iteration of Device Development); Test type: Superiority; p < 0.0001, post-hoc analysis; with Bonferroni correction

5. Primary Outcome: Tidal Volume
Description: as for outcome 4
Time Frame: 10 minutes
Population: Three datasets were discarded due to poor data quality due to instrumentation issues encountered during testing.
Measure: Mean (Standard Error); unit: liters
Arm/Group | Healthy Volunteers (1st Iteration of Device Development)
Number analyzed (Participants) | 16
liters
  Baseline | 0.55 (0.04)
  Vibration | 0.68 (0.09)
Statistical Analysis 1: Comparison: Healthy Volunteers (1st Iteration of Device Development); Test type: Superiority; p = 0.094, post-hoc analysis; with Bonferroni correction

6. Primary Outcome: EMG
Description: Simultaneous multi-frequency synchronous excitation was the stimulus, using 15 Hz at shoulders and 25 Hz at feet. Baseline EMG data were recorded prior to commencement of vibration; a 1 second segment was extracted for post processing. For computing muscle activation during vibration, a 10 second EMG segment was extracted after 1 minute of start of the vibration. Extracted signals were filtered to remove artifacts; similar filtering procedures were carried out for EMG signals recorded during MVIC tests and baseline recording. The root-mean square values of EMG signals of vibration and MVIC were calculated. Normalization to MVIC followed (Vibration EMGRMS)/(MVIC EMGRMS) × 100. Bias calculated using (Filtered EMGRMS @ baseline)/(Unfiltered EMGRMS @ baseline); bias-corrected EMG during vibration computed using (Vibration EMGRMS /Bias). Therefore each muscle site has only 1 reported value, representative of the combined effect of multi-frequency excitation provided at shoulders and feet.
Time Frame: baseline and during intervention (not exceeding 1 minute)
Measure: Mean (Standard Error); unit: percentage of MVC
Arm/Group | Healthy Volunteers (1st Iteration of Device Development)
Number analyzed (Participants) | 19
percentage of MVC
  Baseline bellies of soleus (SO) | 13.10 (1.72)
  During vibration bellies of soleus (SO) | 62.67 (17.42)
  Baseline tibialis anterior (TA) | 5.15 (0.75)
  During vibration tibialis anterior (TA) | 11.59 (2.36)
  Baseline gastroenemius lateralis (GL) | 3.17 (0.24)
  During vibration gastroenemius lateralis (GL) | 7.14 (1.16)
  Baseline vastus medialis (VM) | 5.41 (0.64)
  During vibration vastus medialis (VM) | 8.52 (1.25)
  Baseline vastus lateralis (VL) | 4.33 (0.52)
  During vibration vastus lateralis (VL) | 6.57 (0.73)
  Baselin rectus femoris (RF) | 4.82 (1.56)
  During vibration rectus femoris (RF) | 5.58 (0.51)
  Baseline semitendinosus (ST) | 6.31 (1.97)
  During vibration semitendinosus (ST) | 6.64 (0.95)
  Baseline deltoideus medius | 1.23 (0.13)
  During vibration deltoideus medius | 4.25 (1.05)
Statistical Analysis 1: Comparison: Healthy Volunteers (1st Iteration of Device Development); Comparison of Vibration to Baseline for Muscle bellies of Soleus (SO); Test type: Superiority; p = 0.011, ANOVA — Statistical significance level was set at p <0.05 for all tests
Statistical Analysis 2: Comparison: Healthy Volunteers (1st Iteration of Device Development); Comparison of Vibration to Baseline for tibialis anterior (TA); Test type: Superiority; p = 0.012, ANOVA; Statistical significance level was set at p < 0.05 for all tests
Statistical Analysis 3: Comparison: Healthy Volunteers (1st Iteration of Device Development); Comparison of Vibration to Baseline for gastrocnemius lateralis (GL); Test type: Superiority; p = 0.003, ANOVA — Statistical significance level was set at p < 0.05 for all tests
Statistical Analysis 4: Comparison: Healthy Volunteers (1st Iteration of Device Development); Comparison of Vibration to Baseline for vastus medialis (VM); Test type: Superiority; p < 0.001, ANOVA — Statistical significance level was set at p < 0.05 for all tests
Statistical Analysis 5: Comparison: Healthy Volunteers (1st Iteration of Device Development); Comparison of Vibration to Baseline for vastus lateralis (VL); Test type: Superiority; p < 0.0001, ANOVA — Statistical significance level was set at p < 0.05 for all tests
Statistical Analysis 6: Comparison: Healthy Volunteers (1st Iteration of Device Development); Comparison of Vibration to Baseline for rectus femoris (RF); Test type: Superiority; p = 0.59, ANOVA — Statistical significance level was set at p <0.05 for all tests
Statistical Analysis 7: Comparison: Healthy Volunteers (1st Iteration of Device Development); Comparison of Vibration to Baseline for semitendinosus (ST); Test type: Superiority; p = 0.86, ANOVA — Statistical significance level was set at p < 0.05 for all tests
Statistical Analysis 8: Comparison: Healthy Volunteers (1st Iteration of Device Development); Comparison of Vibration to Baseline for deltoideus medius; Test type: Superiority; p = 0.006, ANOVA — Statistical significance level was set at p < 0.05 for all tests

ADVERSE EVENTS:
Time Frame: AEs were collected only on the days of testing for occurrences during testing sessions. Testing sessions lasted 2-3 hours and the maximum time between first and last session was 146 days, though a more typical spread was 35 days. (Sessions were held at the participant's convenience.)
Arm/Group | Healthy Volunteers (1st Iteration of Device Development)
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Volunteers (1st Iteration of Device Development) (N=22)
Discomfort (General disorders) | 3 — Feeling of unpleasantness, something akin to nausea, but without concern for vomiting

LIMITATIONS AND CAVEATS:
One cannot extrapolate the results of this study to patients at risk for PICS from prolonged immobilization. Study participants were healthy and led relatively active lifestyles. Critically ill and injured patients who are immobilized might not realize physiologic responses similar to or greater than those of this cohort. This study doesn't show whether the degree of muscle activation changes observed with WBV would act as a significant mitigator of atrophy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT03479008/Prot_SAP_000.pdf